CLINICAL TRIAL: NCT06577337
Title: A Phase 1, Randomized, Double-Blind, Sponsor-Open, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Immunogenicity, and Pharmacokinetics of Single Ascending Doses of M5542 Administered Subcutaneously in Healthy Participants
Brief Title: Phase 1 Single Ascending Doses (SAD) of M5542 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: MS201491_0001A; 2024-513069-37-00 (Other: EU CT)
Record Dates: First submitted 2024-08-22; First posted 2024-08-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: First-in-Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M5542 (Experimental)
  Interventions: Biological: M5542
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: M5542 — Participants will receive a single ascending dose of M5542 subcutaneously on Day 1.
  Arms: M5542
Biological: Placebo — Participants will receive a single dose of placebo matched to M5542 subcutaneously on Day 1.
  Arms: Placebo

SUMMARY:
The present study in healthy participants will assess the safety, tolerability, immunogenicity, pharmacokinetics (PK) and pharmacodynamics (PD) of single ascending doses (SAD) of subcutaneously administered M5542.

ELIGIBILITY:
Inclusion Criteria:

* Participants are overtly healthy, as determined by medical evaluation, by physical examination or laboratory evaluation and no active clinically significant disorder, condition, infection, or disease that would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion at Screening and Day -1
* Participants have a body weight within the range 50 to 100 kilograms (kg) (inclusive) and body mass index (BMI) within the range 18 to 30.0 kilograms per square meter kg/m^2 (inclusive) at Screening
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* History or presence of clinically relevant respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, musculoskeletal, genitourinary, immunological, dermatological, connective tissue, psychiatric and other diseases or disorders, and epilepsy, as determined by medical evaluation at Screening and Day -1
* Any condition, including findings in the laboratory tests or other screening assessments, that in the opinion of the Investigator constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study's objectives, conduct, or evaluation at Screening and on Day -1
* History of any malignancy
* History of chronic or recurrent acute infection or any bacterial, viral, parasitic, or fungal infections within 30 days prior to Screening and at any time between Screening and admission, or hospitalization due to infection within 6 months prior to Screening
* Immunization with any vaccine 42 days prior to dosing on Day 1 or planned within 3 months after the last administration of study intervention
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2027-03-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to Day 85
Number of Participants with Abnormal Laboratory Assessments, 12-Lead Electrocardiogram (ECG), and Vital Signs | Up to Day 85

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Serum Concentrations of M5542 | Pre-dose up to 1344 hours post-dose
Number of Participants with Anti-Drug Antibodies (ADA) Against M5542 | Pre-dose up to Day 57

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Clinical Pharmacology Unit of Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201491_0001A
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html